CLINICAL TRIAL: NCT04455581
Title: Open-label, Single-arm, Multicentre Study to Evaluate Efficacy and Safety of SHR-1209 in Subjects With Homozygous Familial Hypercholesterolemia
Brief Title: A Study to Determine the Safety, Tolerability, and Efficacy of SHR-1209 in Patients With Familial Hypercholesterolemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1209-201
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): SHR-1209 administered by subcutaneous injection Atorvastatin or Rosuvastatin combined with Ezetimibe oral
  Interventions: Drug: SHR-1209

INTERVENTIONS:
Drug: SHR-1209 — SHR-1209 administered by subcutaneous injection Atorvastatin or Rosuvastatin combined with Ezetimibe oral

SUMMARY:
The study is being conducted to evaluate the efficacy, safety and tolerability of SHR-1209 in subjects with familial hypercholesterolemia. 8 eligible patients (aged ≥18 years) with familial hypercholesterolemia, on stable maximum tolerable dose lipid-regulating therapy for at least 28 days, to receive subcutaneous SHR-1209, follow up 8 weeks. The primary endpoint was percentage change in LDL cholesterol from baseline at week 12 .

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age
* Diagnosis of homozygous familial hypercholesterolemia
* Stable lipid-lowering therapies for at least 28 days
* LDL cholesterol ≥ 130 mg/dl (3.4 mmol/L)
* Triglyceride ≤ 400 mg/dL (4.5 mmol/L)
* Bodyweight of ≥ 40 kg at screening.

Exclusion Criteria:

* LDL or plasma apheresis within 8 weeks prior to randomization
* New York Heart Association (NYHA) class III or IV or last known left ventricular ejection fraction < 30%
* Myocardial infarction, unstable angina, percutaneous coronary intervention, coronary artery bypass graft or stroke within 3 months of randomization, Planned cardiac surgery or revascularization, Uncontrolled cardiac arrhythmia
* Liver transplant history.
* Uncontrolled hypertension.
* Moderate to severe renal dysfunction.
* Active liver disease or hepatic dysfunction.
* Known sensitivity to any of the products to be administered during dosing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in LDL-C at Week 12 | Week 12

SECONDARY OUTCOMES:
Change From Baseline in LDL-C at Week 12 | Week 12
Percent Change From Baseline in LDL-C at the Mean of Weeks 10 and 12 | Weeks 10 and 12
Change From Baseline in LDL-C at the Mean of Weeks 10 and 12 | Weeks 10 and 12
Percent Change From Baseline in the Total Cholesterol at the Mean of Weeks 10 and 12 | Weeks 10 and 12
Percent Change From Baseline in the Total Cholesterol at Week 12 | Week 12
Percent Change From Baseline in HDL-C at the Mean of Weeks 10 and 12 | Weeks 10 and 12
Percent Change From Baseline in HDL-C at Week 12 | Week 12
Percent Change From Baseline in Non-HDL-C at the Mean of Weeks 10 and 12 | Weeks 10 and 12
Percent Change From Baseline in Non-HDL-C at Week 12 | Week 12
Percent Change From Baseline in Triglycerides at the Mean of Weeks 10 and 12 | Weeks 10 and 12
Percent Change From Baseline in Triglycerides at Week 12 | Week 12
Percent Change From Baseline in Apo B at the Mean of Weeks 10 and 12 | Weeks 10 and 12
Percent Change From Baseline in ApoB at Week 12 | Week 12
Percent Change From Baseline in Apo A1 at the Mean of Weeks 10 and 12 | Weeks 10 and 12
Percent Change From Baseline in Apo A1 at Week 12 | Week 12
Percent Change From Baseline in Lipo(a) at the Mean of Weeks 10 and 12 | Weeks 10 and 12
Percent Change From Baseline in Lipo(a) at Week 12 | Week 12
Number of investigational product-related adverse events | Weeks 12 and 20
Number of ADA and Nab | Week 20

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shu C, Wang Y, Feng S, Yang S, Shen K. Population Pharmacokinetics and Pharmacodynamics Modeling for the Use of Recaticimab in Healthy Volunteers and Patients with Hypercholesterolemia. Clin Pharmacokinet. 2025 Sep;64(9):1341-1355. doi: 10.1007/s40262-025-01512-5. Epub 2025 Jun 30. PMID 40587053